CLINICAL TRIAL: NCT05084482
Title: External Validation of Delirium Prediction Models for Intensive Care Patients. A Prospective, Multicenter, Cohort Study
Brief Title: External Validation of Delirium Prediction Models for Intensive Care Patients
Status: Completed | Type: Observational
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Lone Musaeus Poulsen, Head of ICU, Zealand University Hospital
Other Study IDs: ZUH.01
Record Dates: First submitted 2021-10-06; First posted 2021-10-19 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2023-01

CONDITIONS: Delirium
Keywords: Critical illness; ICU; Delirium; prediction; Observational
MeSH Terms: conditions — Delirium; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients admitted to Intensive Care Unit (ICU): Eligible patients are scored by E-PRE-DELIRIC at admission and PRE-DELIRIC 24 hours after admission.
  Interventions: Other: Prediction models

INTERVENTIONS:
Other: Prediction models — The prediction scores are validated by the CAM-ICU scores up to 14 days after ICU admission.
  Other Names: Delirium; PRE-DELIRIC; E-PRE-DELIRIC

SUMMARY:
Delirium is frequently observed among critically ill patients and is associated with detrimental outcomes. Currently, no evidence-based prevention or treatment exists for delirium, and especially, the inability to identify effective preventive measures of delirium has increased the focus on identifying patients with a high risk of delirium through prediction models. Two prediction models have been developed to estimate the risk of delirium in ICU patients: the prediction model for delirium (PRE-DELIRIC) and the early prediction model for delirium (E-PRE-DELIRIC). These robust and well-calibrated prediction models have the potential of assisting in identifying patients with the highest risk for delirium and thereby to focusing preventive strategies on the most vulnerable group. However further validation is needed in a Danish population.

DETAILED DESCRIPTION:
Adult ICU patients admitted to the participating ICUs in the Region Zealand are included according to eligibility.

Eligible patients will be assessed with E-PREDELIRIC at admission to the ICU and PREDELIRIC 24h after admission to the ICU. Patients will be screened twice daily with CAM-ICU until ICU discharge, death, transferal to non-participating ICU or for a maximum observation period of 14 days.

Central screening via EPIC PDM and registration in central database (REDCap, ZUH) by the principal investigator.

The following are registered: Age, sex, history of cognitive impairment, history of alcohol abuse, admission category, urgent admission, mean arterial blood pressure at the time of ICU admission, use of corticosteroids, respiratory failure, Blood Urea Nitrogen/Carbamide, APACHE-II score, administered morphine does, use of sedatives, metabolic acidosis, coma, presence of infection, delirium status by CAM-ICU, time of ventilation, length of ICU and hospital stay, mortality.

ELIGIBILITY:
Inclusion Criteria:

* Acute admission to an ICU AND
* Age > 18 of years

Exclusion Criteria:

* Total admittance to the ICU less than 24 hours
* Delirium assessment nonapplicable (hearing or visual disabilities, language barriers, or mentally incompetent

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male or female
Study Population: All adult patients admitted to participating ICUs in the Zealand Region between November 2021 and July 2022.
Sampling Method: Non-Probability Sample
Enrollment: 660 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
AUROC for PRE-DELIRIC | Duration of the study, november 2021 to september 2022
  Area Under the Receiver Operating Characteristics (AUROC) for PRE-DELIRIC
AUROC for E-PRE-DELIRIC | Based on 14 days of ICU admission
  Area Under the Receiver Operating Characteristics (AUROC) for E-PRE-DELIRIC

SECONDARY OUTCOMES:
30-days mortality | 30 days efter ICU admission
  Dead or alive at day 30 after ICU admission
Time on ventilator | 14 days after ICU admission
  Days in need of mechanical ventilation up to 14 days of ICU admission
ICU length of stay | 30 days after ICU admission
  Days in the ICU up to 30 days
Hospital length of stay | 30 days after ICU admission
  Days in the hospital up to 30 days after ICU admission

CONTACTS AND LOCATIONS:
Overall Officials: Neeliya Anton Joseph, BSc Medicine, Principal Investigator — Department of Anaesthesiology, Zealand University Hospital, Køge, Denmark
Locations (1):
- Zealand University Hospital, Department of Anaesthesiology, Køge, Zealand Region of Denmark, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Individual anonymised participant data will be made available to researchers upon reasonable request after termination and publication of the study.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After the termination and publication of the study
Access Criteria: Reasonable request by researcher based on study protocol.